CLINICAL TRIAL: NCT01134939
Title: Non-interventional Observational Study With Viramune® Plus Antiretroviral Backbone Combination in HIV-infected Women and Male Patients. Gender Specific Evaluation of Data.
Brief Title: Non-interventional Observational Study With Viramune® in HIV to Evaluate Gender Specific Data
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1536
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- HIV-infected women and men

SUMMARY:
The question that prompted this study is the extent to which results from clinical trials can be translated into everyday practice (external validity). First and foremost are questions about tolerability and the efficacy of an antiretroviral combination treatment with Viramune and other antiretroviral partners. In particular, adverse events will be recorded depending on gender and the therapeutic effect will be monitored via the course of viral load and improvement of the immune system, based on the CD4 cell count.

DETAILED DESCRIPTION:
Time Perspective:

retro- and prospective

ELIGIBILITY:
Inclusion criteria:

The inclusion criteria for treatment with Viramune plus other antiretroviral combination drugs are to be based on the current Information for Healthcare Professionals/SPC

Exclusion criteria:

The inclusion criteria for treatment with Viramune plus other antiretroviral combination drugs are to be based on the current Information for Healthcare Professionals/SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (34):
- Germany (34):
  - Boehringer Ingelheim Investigational Site 23, Aachen
  - Boehringer Ingelheim Investigational Site 10, Berlin
  - Boehringer Ingelheim Investigational Site 11, Berlin
  - Boehringer Ingelheim Investigational Site 14, Berlin
  - Boehringer Ingelheim Investigational Site 19, Berlin
  - Boehringer Ingelheim Investigational Site 26, Berlin
  - Boehringer Ingelheim Investigational Site 28, Berlin
  - Boehringer Ingelheim Investigational Site 33, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site 31, Chemnitz
  - Boehringer Ingelheim Investigational Site 25, Cologne
  - Boehringer Ingelheim Investigational Site 29, Dortmund
  - Boehringer Ingelheim Investigational Site 27, Düsseldorf
  - Boehringer Ingelheim Investigational Site 17, Frankfurt
  - Boehringer Ingelheim Investigational Site 1, Frankfurt
  - Boehringer Ingelheim Investigational Site 2, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 34, Giessen
  - Boehringer Ingelheim Investigational Site 22, Hamburg
  - Boehringer Ingelheim Investigational Site 6, Hamburg
  - Boehringer Ingelheim Investigational Site 12, Hanover
  - Boehringer Ingelheim Investigational Site 16, Hanover
  - Boehringer Ingelheim Investigational Site 32, Karlsruhe
  - Boehringer Ingelheim Investigational Site 15, Koblenz
  - Boehringer Ingelheim Investigational Site 21, Leipzig
  - Boehringer Ingelheim Investigational Site 20, München
  - Boehringer Ingelheim Investigational Site 24, München
  - Boehringer Ingelheim Investigational Site 3, München
  - Boehringer Ingelheim Investigational Site 7, München
  - Boehringer Ingelheim Investigational Site 13, Münster
  - Boehringer Ingelheim Investigational Site 18, Osnabrück
  - Boehringer Ingelheim Investigational Site 30, Stuttgart

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment-naive Female Patients: Female patients who were not pretreated with HIV therapy.
- Treatment-naive Male Patients: Male patients who were not pretreated with HIV therapy.
- Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL: Female patients switching from a virologically effective treatment regimen (i.e. due to intolerance), with a viral load ≤ 50 copies/mL.
- Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL: Male patients switching from a virologically effective treatment regimen (i.e. due to intolerance), with a viral load ≤ 50 copies/mL.
- Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL: Female patients switching from a virologically ineffective treatment regimen, viral load >50 copies/mL.
- Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL: Male patients switching from a virologically ineffective treatment regimen, viral load >50 copies/mL.
- Female Patients, Baseline Viral Load Not Documented: Female patients who could not be assigned to one of the three subgroups and had no documented viral load value.
- Male Patients, Baseline Viral Load Not Documented: Male patients who could not be assigned to one of the three subgroups and had no documented viral load value.
Period: Overall Study
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Started | 59 | 42 | 51 | 46 | 33 | 14 | 19 | 1
Completed | 42 | 24 | 41 | 32 | 23 | 5 | 10 | 1
Not Completed | 17 | 18 | 10 | 14 | 10 | 9 | 9 | 0
Not completed — Adverse Event | 9 | 3 | 4 | 5 | 5 | 5 | 1 | 0
Not completed — Lack of Efficacy | 2 | 5 | 1 | 0 | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Termination page not available | 4 | 6 | 5 | 8 | 0 | 3 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set includes all HIV-1 infected patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment and of an antiretroviral combination partner.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented | Total
Number analyzed (Participants) | 59 | 42 | 51 | 46 | 33 | 14 | 19 | 1 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.7) | 39.2 (11.2) | 39.2 (9.1) | 44.2 (8.1) | 36.3 (8.0) | 43.2 (10.7) | 38.9 (8.9) | 50.0 | 39.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 0 | 51 | 0 | 33 | 0 | 19 | 0 | 162
  Male | 0 | 42 | 0 | 46 | 0 | 14 | 0 | 1 | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Virologic Response (VR) After 36 Months
Description: VR is defined as HIV viral load of < 50 copies/mL before month 36 and without subsequent rebound or change of ARV therapy. A rebound is defined by two consecutive measurements of VL ≥ 50 copies/ml, at least two weeks apart.
  A change of ARV therapy is defined as a permanent discontinuation of Viramune®. A change in the background therapy due to toxicity or intolerance is not considered failure for the analysis. Therefore, a patient remains a treatment responder in this case if all other criteria are fulfilled. A rebound is defined by two consecutive measurements of VL ≥ 50 copies/ml, at least two weeks apart, after two consecutive measurements of VL< 50 copies/ml.
Time Frame: 36 months
Population: Patients from Full Analysis Set (FAS): This patient set includes all patients in the treated set who have analysable data in at least one efficacy endpoint.
Measure: Number; unit: participants
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 58 | 42 | 51 | 46 | 33 | 14 | 18 | 1
participants | 44 | 30 | 46 | 40 | 25 | 6 | 16 | 1

2. Secondary Outcome: Changes in the Viral Load After 36 Months From Baseline
Description: The change in the log10 viral load from baseline after 36 months was calculated by subtracting the baseline value from the value after 36 months. Therefore, a negative change represents a decrease in viral load.
Time Frame: Baseline and 36 months
Population: Patients from FAS with values for viral load at baseline and after 36 months.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 45 | 36 | 51 | 45 | 30 | 12 | 0 | 0
Log10 copies/mL | -2.7 (1.2) | -2.7 (1.5) | -0.3 (0.7) | -0.3 (0.5) | -2.4 (1.7) | -1.2 (1.3) |  |

3. Secondary Outcome: Changes in the CD4+ Cell Count After 36 Months From Baseline
Description: The change in the Cluster of differentiation 4 (CD4+) cell count from baseline after 36 months was calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase in CD4+ cell count.
Time Frame: Baseline and 36 months
Population: Patients from FAS with values for CD4+ at baseline and after 36 months.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 44 | 35 | 50 | 45 | 30 | 12 | 1 | 1
cells/mm^3 | 253.3 (209.9) | 216.9 (191.4) | 85.9 (196.6) | 39.8 (193.6) | 246.4 (271.2) | 137.1 (301.8) | 115.0 | 342.0

4. Secondary Outcome: Changes in the Laboratory Data (Total Cholesterol) After 36 Months From Baseline
Description: The changes in the laboratory data (Total Cholesterol) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for total cholesterol at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 14 | 5 | 9 | 5 | 13 | 1 | 2 | 0
mg/dL | 3.9 (61.0) | 32.9 (20.8) | -11.5 (60.3) | 43.0 (37.6) | -2.0 (34.5) | 26.0 (NA) — N=1 | 74.0 (32.5) |

5. Secondary Outcome: Changes in the Laboratory Data (HDL Cholesterol) After 36 Months From Baseline
Description: The changes in the laboratory data ( High density protein (HDL) Cholesterol) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for HDL cholesterol at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 7 | 3 | 6 | 5 | 6 | 0 | 2 | 0
mg/dL | 15.6 (15.5) | 20.2 (1.0) | 9.3 (17.1) | -26.5 (102.8) | 18.9 (13.1) |  | 5.0 (21.2) |

6. Secondary Outcome: Changes in the Laboratory Data (LDL Cholesterol) After 36 Months From Baseline
Description: The changes in the laboratory data (Low density protein (LDL) Cholesterol) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for LDL cholesterol at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 7 | 3 | 6 | 5 | 6 | 0 | 2 | 0
mg/dL | 5.3 (30.3) | 27.8 (13.9) | 3.8 (24.3) | 5.0 (30.4) | -9.3 (27.8) |  | 73.0 (42.4) |

7. Secondary Outcome: Changes in the Laboratory Data (Triglycerides) After 36 Months From Baseline
Description: The changes in the laboratory data (Triglycerides) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for triglycerides at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 14 | 5 | 9 | 6 | 13 | 1 | 2 | 0
mg/dL | -18.5 (63.1) | -16.6 (32.3) | -71.8 (102.2) | -31.7 (90.8) | -53.3 (53.7) | 160 (NA) — N=1 | -5.5 (50.2) |

8. Secondary Outcome: Changes in the Laboratory Data (Blood Glucose) After 36 Months From Baseline
Description: The changes in the laboratory data (Blood Glucose) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for blood glucose at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 14 | 5 | 11 | 4 | 15 | 1 | 3 | 0
mg/dL | 2.4 (29.1) | 5.3 (18.6) | 0.2 (22.2) | 3.9 (7.2) | 7.2 (13.8) | -27.5 (NA) — N=1 | -17.3 (38.5) |

9. Secondary Outcome: Changes in the Laboratory Data ( ALT) After 36 Months From Baseline
Description: The changes in the laboratory data (Alanine transaminase (ALT)) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for ALT at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 13 | 7 | 9 | 9 | 16 | 2 | 3 | 0
U/L | 1.3 (8.6) | 7.5 (13.8) | 7.7 (11.7) | 6.1 (18.7) | 0.0 (15.4) | 12.6 (34.8) | 6.3 (11.7) |

10. Secondary Outcome: Changes in the Laboratory Data (AST) After 36 Months From Baseline
Description: The changes in the laboratory data (Aspartate transminase (AST)) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for the AST at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 13 | 7 | 8 | 9 | 16 | 2 | 3 | 0
U/L | 1.4 (9.5) | 3.0 (11.2) | 1.4 (5.6) | 0.4 (10.3) | -1.7 (13.5) | -0.8 (17.3) | 0.7 (6.1) |

11. Secondary Outcome: Changes in the Laboratory Data (Gamma-GT) After 36 Months From Baseline
Description: The changes in the laboratory data (Gamma glutamyl transferase (Gamma GT)) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Gamma GT at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 14 | 7 | 9 | 9 | 16 | 2 | 3 | 0
U/L | 22.7 (26.9) | 25.2 (15.4) | 7.0 (25.7) | 4.8 (111.7) | 20.9 (31.6) | 40.8 (61.9) | -4.7 (10.5) |

12. Secondary Outcome: Changes in the Laboratory Data (Creatinine) After 36 Months From Baseline
Description: The changes in the laboratory data (Creatinine) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for creatinine at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 13 | 7 | 10 | 9 | 16 | 2 | 3 | 0
mg/dL | 0.0 (0.2) | 0.1 (0.1) | -0.1 (0.2) | -0.1 (0.1) | 0.0 (0.1) | -0.1 (0.0) | 0.0 (0.1) |

13. Secondary Outcome: Changes in the Laboratory Data (Haemoglobin) After 36 Months From Baseline
Description: The changes in the laboratory data (Haemoglobin) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data. .
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for haemoglobin at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment-naive Female Patients | Treatment-naive Male Patients | Pretreated Female Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Female Patients, Baseline Viral Load > 50 Copies/mL | Pretreated Male Patients, Baseline Viral Load > 50 Copies/mL | Female Patients, Baseline Viral Load Not Documented | Male Patients, Baseline Viral Load Not Documented
Number analyzed (Participants) | 14 | 7 | 9 | 9 | 16 | 2 | 3 | 0
g/dL | 0.8 (1.3) | 0.4 (0.8) | 0.1 (1.1) | 0.8 (1.0) | 1.1 (1.1) | 1.0 (2.4) | 0.3 (1.8) |

ADVERSE EVENTS:
Time Frame: 36 months
Groups:
- Treatment-naive Patients: Female and male patients who were not pretreated with HIV therapy.
- Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL: Female and male patients switching from a virologically effective treatment regimen (i.e. due to intolerance), with a viral load ≤ 50 copies/mL.
- Pretreated Patients, Baseline Viral Load > 50 Copies/mL: Female and male patients switching from a virologically ineffective treatment regimen, viral load >50 copies/mL.
- Patients With Baseline Viral Load Not Documented: Female and male patients who could not be assigned to one of the three subgroups and had no documented viral load value.
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Serious Adverse Events (participants affected / at risk) | 7/101 | 10/97 | 4/47 | 1/20
Other Adverse Events (participants affected / at risk) | 46/101 | 56/97 | 24/47 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naive Patients (N=101) | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL (N=97) | Pretreated Patients, Baseline Viral Load > 50 Copies/mL (N=47) | Patients With Baseline Viral Load Not Documented (N=20)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster infection neurological (Infections and infestations) | 0 | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naive Patients (N=101) | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL (N=97) | Pretreated Patients, Baseline Viral Load > 50 Copies/mL (N=47) | Patients With Baseline Viral Load Not Documented (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 11 | 3 | 2
Nausea (Gastrointestinal disorders) | 11 | 7 | 3 | 2
Asthenia (General disorders) | 3 | 6 | 2 | 1
Fatigue (General disorders) | 9 | 9 | 2 | 1
Bronchitis (Infections and infestations) | 10 | 13 | 5 | 1
Gastroenteritis (Infections and infestations) | 2 | 3 | 4 | 1
Herpes zoster (Infections and infestations) | 4 | 1 | 3 | 1
Infection (Infections and infestations) | 5 | 7 | 2 | 1
Nasopharyngitis (Infections and infestations) | 5 | 6 | 4 | 2
Sinusitis (Infections and infestations) | 3 | 4 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 12 | 12 | 8 | 3
Urinary tract infection (Infections and infestations) | 2 | 6 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 6 | 2 | 0
Blood cholesterol increased (Investigations) | 5 | 6 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 8 | 16 | 6 | 1
Low density lipoprotein increased (Investigations) | 4 | 5 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 5 | 1 | 0
Headache (Nervous system disorders) | 7 | 11 | 4 | 3
Depression (Psychiatric disorders) | 3 | 15 | 3 | 1
Sleep disorder (Psychiatric disorders) | 3 | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.